CLINICAL TRIAL: NCT01741168
Title: TLSO Versus No Orthosis for the Treatment of Thoracolumbar Burst Fractures Without Neurologic Injury: A Multicenter Prospective Randomized Equivalence Trial
Brief Title: Brace Versus No Brace for the Treatment of Thoracolumbar Burst Fractures Without Neurologic Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The London Spine Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11421
Record Dates: First submitted 2012-11-22; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Thoracolumbar Burst Fractures Without Neurologic Deficit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TLSO (Active Comparator): TLSO brace 8-10 weeks
  Interventions: Other: TLSO
- No Orthosis (Experimental): No Orthosis
  Interventions: Other: No Orthosis

INTERVENTIONS:
Other: TLSO — Patients in the TLSO arm will remain on bed rest until fitted with a TLSO. They will wear the TLSO for 8-10 weeks and mobilized in the brace by a physiotherapist.
  Other Names: TLSO Aspen Medical Products, Irvine, CA, USA
  Arms: TLSO
Other: No Orthosis — Patients in the No Orthosis group will be mobilized immediately as tolerated by a physiotherapist with restrictions to limit bending or rotating through their trunk. They will be encouraged to return to normal activities after 8 weeks.
  Arms: No Orthosis

SUMMARY:
Braces have been used o treat stable (not requiring surgery) burst fractures with much success. Recently questions have been raised in regards to the importance of the brace. Some studies have results that suggest a brace is not important in having a good outcome. However, this has never been proven. This study is being conducted to see whether or not wearing a brace is important to having a good outcome.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively compare the outcome between patients randomly assigned to a thoracolumbosacral orthosis (TLSO) treatment group or no orthosis (NO) treatment group, for the management of an acute AO type A3 thoracolumbar fracture.

ELIGIBILITY:
Inclusion Criteria:

* AO A3 burst fracture between T10 and L3 with associated kyphotic deformity <35 degrees
* neurologically intact or isolated nerve root deficit
* age 16-60 years
* enrollment within 3 days of injury

Exclusion Criteria:

* neurological deficit
* can not comply with brace wearing (pregnancy/body mass index >40)
* mobilized with or without a brace prior to recruitment
* suffered a pathologic or open fracture
* alcohol or drug abusers
* had previous injury or surgery to the thoracolumbar region
* unable to complete the questionnaires

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2005-06; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | 3 months post fracture
  The primary outcome measure is the Roland Morris Disability Questionnaire (RMDQ) administered at 3 months post fracture. The RMDQ evaluates physical disability secondary to low back pain and is validated, simple to administer, sensitive, and reliable. The questionnaire evaluates 24 items to derive a score that varies between zero (no disability) and twenty-four (severe disability). Three months was chosen because it is the time point at which we expect a significant functional recovery and readiness to resume most normal activities.

SECONDARY OUTCOMES:
SF-36 physical component summary score | enrollment, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2years
SF-36 mental component summary score | enrollment, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
VAS pain score | enrollment, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
Satisfaction with Treatment | enrollment, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  Overall satisfaction with treatment was assessed on a seven point scale, using the sentence, "All things considered, how satisfied are you with the results of your recent treatment for your spine fracture?" This is a recommended tool for assessing global satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- London Spine Centre, London, Ontario, Canada